CLINICAL TRIAL: NCT00518973
Title: Double-blind Placebo-controlled Trial of Quetiapine in Anorexia Nervosa
Brief Title: Trial of Quetiapine in Anorexia Nervosa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of South Florida (Other)
Responsible Party: Principal Investigator, Walter Kaye, Program Director and Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 051027; QUET0376
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Results first posted 2019-07-17 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-06

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): The primary outcome was to determine the effect of quetiapine compared with placebo in terms of reducing core eating disorder symptoms on the Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS) and the Eating Disorder Inventory-2 (EDI-2).
  Interventions: Drug: Placebo
- Quetiapine (Experimental): Secondary outcomes were to determine if quetiapine is superior to placebo in reducing anxiety, depression and obsessionality assessed with the State Trait Anxiety Inventory (STAI), Hamilton Depression Rating Scale (HAM D) and Yale-Brown Obsessive Compulsive Scale, respectively. In addition, another secondary goal was to determine if quetiapine is superior to placebo in terms of weight gain. Adverse events were also determined.
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Quetiapine — Subjects will start with 25mg hs on day 1, 25mg bid on day 2, 25mg am and 50mg hs on day 3, 50mg bid on day 4, 50mg am and 75mg hs on day five, and 75mg bid on day six. Dosage will be increased further on an individual basis as determined by the study physician and as tolerated by the subject with a maximum dosage of 400 mg. Dose can be reduced as determined by clinical judgment. In order to determine the most effective dose, the dose of Quetiapine (or placebo) will be titrated at intervals by staff according to the previously stated guidelines, the Pittsburgh Quetiapine Medication Management Assessment and Interview. Subjects will be interviewed about the factors described above and medication dose will be adjusted upward or downward depending upon symptom persistence or side effects.
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Placebo — Subjects will start with 25mg hs on day 1, 25mg bid on day 2, 25mg am and 50mg hs on day 3, 50mg bid on day 4, 50mg am and 75mg hs on day five, and 75mg bid on day six. Dosage will be increased further on an individual basis as determined by the study physician and as tolerated by the subject with a maximum dosage of 400 mg. Dose can be reduced as determined by clinical judgment. In order to determine the most effective dose, the dose of placebo will be titrated at intervals by staff according to the previously stated guidelines, the Pittsburgh Quetiapine Medication Management Assessment and Interview. Subjects will be interviewed about the factors described above and medication dose will be adjusted upward or downward depending upon symptom persistence or side effects.
  Arms: Placebo

SUMMARY:
This research study is being held at UCSD to determine whether the medication Quetiapine helps people suffering from anorexia nervosa by reducing core eating disorders symptoms. This study will see if the medication Quetiapine helps symptoms of anxiety, depression, and obsessionality, in addition to increasing BMI. Men and women between the ages of 18-65 and are currently suffering from anorexia nervosa are needed.

ELIGIBILITY:
Inclusion Criteria:

* Meet criteria for DSM-IV anorexia nervosa (restricting or binge-eating/purging types)
* At least 15% below ideal body weight
* Judged to be reliable to keep clinic visits and able to take all tests and examinations required by the protocol and be able to understand and decide whether or not to sign the Informed Consent.

Exclusion Criteria:

Subjects will not be included in the study who present with any of the following:

* Schizophrenia or schizoaffective disorder (DSM-IV)
* Any ECG abnormality considered clinically significant by the investigator
* Subjects with liver enzymes elevated two times or more above normal
* Other laboratory abnormalities considered clinically significant by the investigator including laboratory deviations requiring acute medical intervention
* Pregnant women, women of childbearing potential not using medically accepted means of contraception (abstinence, IUD, birth control pills, barrier devices or implanted progesterone rods stabilized for at least three months), and lactating women
* Serious suicide risk
* Any medical condition that would preclude the outpatient treatment of anorexia nervosa or the use of quetiapine
* Organic brain disease
* History of severe allergies
* Multiple adverse drug reactions or known allergy to quetiapine
* Use of neuroleptic medications (except benzodiazepines) within 7 days preceding randomization
* History of alcohol or substance abuse disorder as defined in the DSM-IV within the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Kaye, MD, Principal Investigator — University of California, San Diego and University of Pittsburg
Locations (1):
- UCSD Department of Psychiatry Center for Eating Disorder Research, San Diego, California, United States

REFERENCES:
- [Result] Powers PS, Klabunde M, Kaye W. Double-blind placebo-controlled trial of quetiapine in anorexia nervosa. Eur Eat Disord Rev. 2012 Jul;20(4):331-4. doi: 10.1002/erv.2169. Epub 2012 Apr 26. PMID 22535517

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of these 21, 15 were randomized and began the drug; the other six participants failed the in-person screening phase.
Period: Overall Study
Arm/Group | Placebo | Quetiapine
Started | 9 | 6
Completed | 6 | 4
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The data is not available | NA (NA) — The data is not available | 34 (13.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not available | NA — Data not available | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not available | NA — Data not available | NA — Total not calculated because data are not available (NA) in one or more arms.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Hours Occupied by Preoccupations and Rituals Assessed by Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS)
Description: The YBC-EDS is an eight-item scale assessing severity of preoccupations and rituals.
Time Frame: Day 1 to LOCF (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 9 | 6
Hours
  Hours occupied by preoccupations | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
  Hours occupied by rituals | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .15, t-test, 2 sided — t = 2.8; Hours occupied by preoccupations
Statistical Analysis 2: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .40, t-test, 2 sided — t = .56; Hours of rituals

2. Primary Outcome: Difference in Scores on the EDI-2 (Eating Disorders Inventory)
Description: The EDI consists of 8 subscales measuring drive for thinness, bulimia, body dissatisfaction, ineffectiveness, perfectionism, interpersonal distrust, interoceptive awareness, and maturity fears
Time Frame: Day 1 to LOCF (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 9 | 6
Units on the scale | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .72, t-test, 2 sided — t = .13

3. Secondary Outcome: Difference in Scores on the STAI (State-Trait Anxiety Inventory)
Description: The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety.
Time Frame: Day 1 to LOCF (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 9 | 6
Units on the scale
  Trait | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
  State | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .48, t-test, 2 sided — t = .52; Reporting for Trait
Statistical Analysis 2: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .77, t-test, 2 sided — t = .09; Reporting for State

4. Secondary Outcome: Differences in Scores on the HAM-D (Hamilton Depression Rating Scale)
Description: Hamilton Depression Rating Scale (HAM-D) form lists 21 items, the scoring is based on the first 17. It generally takes 15-20 minutes to complete the interview and score the results. Eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2.
Time Frame: Day 1 to LOCF (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 9 | 6
Units on the scale | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .83, t-test, 2 sided — t = .05

5. Secondary Outcome: Differences in Scores on the PANNSS (The Positive and Negative Syndrome Scale)
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. A clinical interview is conducted and patient is rated from 1 to 7 on 30 different symptoms based on the interview.
Time Frame: Day 1 to LOCF (up to 8 weeks)
Measure: Mean (Standard Deviation); unit: Units on the scale
Arm/Group | Placebo | Quetiapine
Number analyzed (Participants) | 9 | 6
Units on the scale
  Positive Scale | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
  Negative Scale | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
  General Scale | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available. | NA (NA) — Access to raw data is not available, only the statistical analysis from the publication are available.
Statistical Analysis 1: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .40, t-test, 2 sided — t = .78; Positive Scale
Statistical Analysis 2: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .11, t-test, 2 sided — t=3.0; Negative Scale
Statistical Analysis 3: Comparison: Placebo vs Quetiapine; Test type: Superiority; p = .90, t-test, 2 sided — t = .02; General Scale

ADVERSE EVENTS:
Arm/Group | Placebo | Quetiapine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | Quetiapine (N=6)
Worsening weight loss (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Participant was hospitalized for worsening weight loss
Car Accident (Social circumstances) | 0 (0) | 1 (1) — Participant was hospitalized after she was hit by a car while riding a bicycle.
Worsening Manic Symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — Participant was hospitalized for worsening manic symptoms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes